CLINICAL TRIAL: NCT07051733
Title: The Preliminary Effect of a Health Information Literacy Enhancement Program for Community-dwelling Individuals With Metabolic Syndrome: A Feasibility Study Based on the Health Empowerment Theory
Brief Title: Preliminary Effect of a Health Information Literacy Enhancement Program for Individuals With Metabolic Syndrome
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Meihua Ji (Other)
Collaborators: The Luhe Teaching Hospital of the Capital Medical University (Other)
Responsible Party: Sponsor-Investigator, Meihua Ji, Associate Professor, Capital Medical University
Organization: Capital Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Z2023SY119
Record Dates: First submitted 2025-06-02; First posted 2025-07-04 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Metabolic Syndrome (MetS)
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health Information Literacy Enhancement Group (Experimental): A 6-week intervention programme was implemented for the health information literacy enhancement group, once a week, with each intervention lasting 30-40min, to enable the study participants to actively practice healthy behaviours through intervention techniques such as health awareness awakening, social resource building, and health-related skill empowerment, in order to enhance the health information literacy of the study participants, and ultimately to enable the study participants to perceive health in a programmatic manner.
  Interventions: Behavioral: Health Information Literacy Enhancement

INTERVENTIONS:
Behavioral: Health Information Literacy Enhancement — Participants will undertake a six-week programme to enhance their health information literacy. The specific details are as follows:
  1. Capacity Building on Health Information Management via Health Education Based on the Health Empowerment Theory: ① Strengthening skills related to Health Information Literacy; ② Training on Medication Management Skills; ③ Practice of Self-Monitoring Skills; ④ Education on Diet and Exercise Management Knowledge.
  2. Health Behavior Motivation Management Based on the Health Empowerment Theory: ① Personalized Goal Setting; ② Behavioral Incentives and Feedback; ③ Construction of Peer Support Networks; ④ Demonstration Effect of Role Models.
  3. Health Management Support System Based on the Health Empowerment Theory: ① Online Dynamic Monitoring; ② Family-Community Collaborative Support; ③ Digital Monitoring Platform; ④ Continuous Supply of Resources.

SUMMARY:
The purpose of this study is to evaluate the preliminary effect of a health-information literacy promotion program for individuals with Metabolic Syndrome (including its subtypes) based on the Health Empowerment Theory. The study aims to answer the following questions:

Does the intervention improve health information literacy among study participants? Does the intervention lead to better health outcomes, including weight, waist circumference, BMI control, and metabolic health indicators (blood pressure, blood glucose, glycated hemoglobin, and blood lipids)?

Participants will:

Undergo the intervention program for 6 weeks (face to face and online) and will be assessed regularly to monitor changes in their health information literacy and health outcomes.

DETAILED DESCRIPTION:
1. Health information management ability education based on health empowerment theory: ① health information literacy intensive training; ② medication management skills training; ③ self-monitoring skills practice; ④ diet and exercise management knowledge education.
2. Health behaviour motivation management based on health empowerment theory: ① personalized goal setting: set learning goals with patients and clarify the weekly health information literacy improvement plan; ② peer support network construction: set up a discussion group to encourage patients to share their experiences in diet management and exercise practice, and enhance their knowledge of diet and exercise through group interaction; ③ Role model demonstration effect: patients with high health information literacy and remarkable self-management effects are set up as role models, and are invited to share their success stories.
3. Health management support system based on the theory of health empowerment: ① online dynamic supervision: weekly Q&A sessions through WeChat groups to address issues such as health information screening, medication use, and interpretation of monitoring data; ② collaborative family-community support: inviting family members to join the health management group to assist in dietary planning, supervise the implementation of exercise, and linking with the community health service centres to provide personalized guidance; ③ digital monitoring platforms Digital monitoring platform: Using the Concordia Medical Weight Loss applet and diet management WeChat group to push customised health advice; ④Continuous supply of resources: Regularly updating links to authoritative channels, such as the website of the State Drug Administration and the China Public Health Network, to ensure that patients have access to reliable health information.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Patients diagnosed with metabolic syndrome (meeting ≥3 criteria):
* Waist circumference ≥ 90 cm (men) / ≥ 85 cm (women)
* Fasting glucose ≥ 6.1 mmol/L or OGTT 2h-glucose ≥ 7.8 mmol/L and/or diabetes treatment
* Blood pressure ≥ 130/85 mmHg and/or hypertension treatment
* Fasting triglycerides (TG) ≥ 1.70 mmol/L
* Fasting HDL-C < 1.04 mmol/L
* Individuals with ≥1 metabolic abnormality not meeting full metabolic syndrome criteria
* Cognitively aware with literacy skills and voluntary participation

Exclusion Criteria:

* Severe hepatic/renal dysfunction, cancer, or life-threatening diseases
* Mental disorders, visual/hearing impairments, or intellectual disabilities

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-08 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Health Information Literacy | Measurements will be taken once before the formal intervention and once after the intervention ends (at 6 weeks).
  Health information literacy (HIL) is essential to assist individuals in health decision-making. In this study, health information literacy will be measured using the Health Information Literacy Self-rating Scale.A 5-point Likert scale was used, with scores ranging from 1-5 for 'strongly disagree' to 'strongly agree', and a total scale score ranging from 29-145, with higher scores indicating higher levels of health information literacy. In the original study, the Cronbach's α coefficient for HILSS was 0.847, and the Cronbach's α coefficients for the dimensions.

SECONDARY OUTCOMES:
Health Literacy | Measurements will be taken once before the formal intervention and once after the intervention ends (at 6 weeks).
  Health literacy refers to an individual's ability to obtain, process, and understand basic health information and services, and to make appropriate health decisions. Compared with health information literacy, the concept and scope of health literacy are more general and broader. In this study, the Newest Vital Sign scale will be used to assess individuals' overall health literacy levels.The measure has six questions assessing a person's reading, numeracy, and comprehension based on an ice cream nutritional label.1 point for each correct answer, 6 questions in total, total score 0-6 points, the higher the score the higher the health literacy. The internal consistency (Cronbach's α) was 0.76.
Chronic Patient Self-Management Questionnaire | Measurements will be taken once before the formal intervention and once after the intervention ends (at 6 weeks)
  The Self-Management Questionnaire for Chronic Patients used to assess the self-management level of patients with chronic diseases. The scale includes five aspects: dietary habits, exercise management, medication adherence, emotional management, and family and social support, and adopts the Likert 5-point rating method. The questionnaire consists of 20 multiple choice questions with a total score of 100 points. The scoring criteria are: between 20 and 60 points is a poor level of self-management; between 60 and 80 points is a medium level of management; between 80 and 100 points is a high level of self-management. The Cronbach's α coefficient of the scale is 0.957.
Health Problem-Solving | Measurements will be taken once before the formal intervention and once after the intervention ends (at 6 weeks)
  The Chinese version of the Health Problem-Solving Scale consists of 6 dimensions: rational/effective problem-solving, positive positive transfer problem-solving, avoidance problem-solving, impulsive/careless problem-solving, negative transfer/learning, and negative motivation/attitude. It includes 30 items. The Likert 5-point scoring method was used, with the lowest score being 0 and the highest score being 4. The higher the score, the better the health problem solving ability. The content validity index of the scale is 0.970, the content validity index of the items ranges from 0.830 to 1.000, the Cronbach's α coefficient is 0.911, and the Cronbach's α coefficients of each dimension range from 0.715 to 0.839.
Chronic Illness Resources | Measurements will be taken once before the formal intervention and once after the intervention ends (at 6 weeks)
  The Chronic Illness Resource Survey (CIRS) consists of 19 items measuring six aspects of social resources: individuals, family and friends, healthcare team, community, media policy and community organisations. The scale is scored on a 5-point Likert scale, ranging from 1 to 5. Higher scores indicate greater access to or use of resources. The scale had good reliability in the original study, with a Cronbach's α coefficient of 0.820, and an overall Cronbach's α coefficient of 0.845 in the Chinese population.
Health-related Quality of Life | Measurements will be taken once before the formal intervention and once after the intervention ends (at 6 weeks)
  A health-related quality of life scale, the EQ-5D-5L, developed by the EuroQol Group, will be used to measure individuals' quality of life. It comprises the EQ-5D descriptive system and the EQ-5D Visual Analog Scale (EQ VAS). The five dimensions assess participants' mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, with each dimension having five levels: no difficulties, slight difficulties, moderate difficulties, severe difficulties, and extreme difficulties/unable to perform. the UI scores ranged from -0.391 to 1.The EQ VAS records a participant's self-assessed health status on a vertical visual analogue scale labelled 'Your best imagined health (100 points)' and 'Your worst imagined health (0 points)'. The EQ VAS provides a quantitative description of the respondent's perception of their overall health. Higher scores indicate higher quality of life. EQ-5D-5L has been validated by Chinese scholars with a Cronbach coefficient of 0.624.
Nutrition Literacy | Measurements will be taken once before the formal intervention and once after the intervention ends (at 6 weeks)
  The Food and Nutrition Literacy Questionnaire, developed by the School of Public Health at Peking University, will be used for assessment. The current status of nutrition literacy includes four dimensions: knowledge and concepts related to food, selecting food, preparing food, and consuming food. The questionnaire has a score of 100 points, and the critical value of this questionnaire is 80 points, and a score of 80 points or more represents nutritional literacy, and the proportion of patients with nutritional literacy is the level of nutritional literacy. The Cronbach'sａcoefficient of the scale is 0.893, and the content validity is 0.891, which is considered to be good.

CONTACTS AND LOCATIONS:
Overall Officials: Meihua Ji, PhD, Principal Investigator — Capital Medical University School of Nursing
Locations (1):
- Li Yuan Community Health Service Center in Tongzhou District, Beijing, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zhang Y, Zhang Z, Xu M, Aihemaitijiang S, Ye C, Zhu W, Ma G. Development and Validation of a Food and Nutrition Literacy Questionnaire for Chinese Adults. Nutrients. 2022 May 5;14(9):1933. doi: 10.3390/nu14091933. PMID 35565900
- [Result] Hill-Briggs F, Gemmell L, Kulkarni B, Klick B, Brancati FL. Associations of patient health-related problem solving with disease control, emergency department visits, and hospitalizations in HIV and diabetes clinic samples. J Gen Intern Med. 2007 May;22(5):649-54. doi: 10.1007/s11606-006-0091-2. PMID 17443373
- [Result] Glasgow RE, Toobert DJ, Barrera M Jr, Strycker LA. The Chronic Illness Resources Survey: cross-validation and sensitivity to intervention. Health Educ Res. 2005 Aug;20(4):402-9. doi: 10.1093/her/cyg140. Epub 2004 Nov 30. PMID 15572438
- [Result] Luo N, Liu G, Li M, Guan H, Jin X, Rand-Hendriksen K. Estimating an EQ-5D-5L Value Set for China. Value Health. 2017 Apr;20(4):662-669. doi: 10.1016/j.jval.2016.11.016. Epub 2017 Feb 9. PMID 28408009
- [Result] Weiss BD, Mays MZ, Martz W, Castro KM, DeWalt DA, Pignone MP, Mockbee J, Hale FA. Quick assessment of literacy in primary care: the newest vital sign. Ann Fam Med. 2005 Nov-Dec;3(6):514-22. doi: 10.1370/afm.405. PMID 16338915

DOCUMENTS (1):
  • Informed Consent Form (2025-05-01): https://cdn.clinicaltrials.gov/large-docs/33/NCT07051733/ICF_001.pdf